CLINICAL TRIAL: NCT00865462
Title: A Randomized, Single Dose Two -Way Crossover Relative Bioavailability Study of Bupropion XL Tablets Formulation in Normal, Healthy Man Following a Standard Meal
Brief Title: A Relative Bioavailability Study of Bupropion XL 150 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 04-0646-004
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Bupropion; Healthy subjects
MeSH Terms: interventions — Bupropion; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Abrika Bupropion 150 mg XL Tablet, single dose
  Interventions: Drug: Abrika Bupropion 150 mg XL Tablet, single dose
- B (Active Comparator): Wellbutrin XL® 150 mg Tablet, single dose
  Interventions: Drug: Wellbutrin XL® 150 mg Tablet, single dose

INTERVENTIONS:
Drug: Abrika Bupropion 150 mg XL Tablet, single dose — A: Experimental Subjects received Abrika formulated products under fed conditions
  Other Names: Bupropion
  Arms: A
Drug: Wellbutrin XL® 150 mg Tablet, single dose — B: Active comparator Subjects received GlaxoSmithKline formulated products under fed conditions
  Other Names: Bupropion
  Arms: B

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of Abrika Bupropion 150 mg XL Tablet to that of Wellbutrin XL® 150 mg Tablet after a single, one-tablet dose in subjects fed a standard meal.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: A Randomized, Single Dose Two -Way Crossover Relative Bioavailability Study of Bupropion XL Tablets Formulation in Normal, Healthy Man Following a Standard Meal

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Is the individual a healthy, normal adult man who volunteers to participate?
* Is he 18-45 years of age, inclusive?
* Is his BMI ≤30?
* Is he considered reliable and capable of understanding his responsibility and role in the study?
* Has he provided written informed consent? A no answer to any of the above questions indicates that the individual is ineligible for enrollment

Exclusion Criteria:

* Does the individual have a history of allergy or hypersensitivity to bupropion, milk or eggs?
* Does he smoke more than 25 cigarettes/day?
* Is he unable to refrain from smoking during the period beginning two hours before and ending four hours after study drug administration?
* Does he have a history of seizure, cranial trauma, or other predisposition to seizure?
* Does he have clinically significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize his safety?
* Does he have significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hematopoietic, hepatic, neurological, ongoing infection, pancreatic, renal or other diseases, conditions or surgeries that would interfere with the conduct or interpretation of the study or jeopardize his safety?
* Does he have serious psychological illness?
* Does he have significant history (within the past six months) or clinical evidence of alcohol or drug abuse?
* Does he have a positive urine drug screen or saliva alcohol screen, or a positive HIV-l, or hepatitis B or C screen?
* Is he unable to refrain from the use of alcohol or xanthine-containing foods or beverages during periods beginning 24 and 48 hours, respectively, prior to study drug administration and ending when the last blood sample has been taken?
* Has he used any prescription drug during the 14-day period prior to study initiation (except for topical products without systemic absorption), or any OTC drug during the 72-hour period preceding study initiation?
* Is he unable to refrain from the use of all concomitant medications during the study?
* Has he donated or lost blood, or participated in a clinical study which involved the withdrawal of a large volume of blood (480 mL or more), during the six week period preceding study initiation?
* Has he donated plasma during the two week period preceding study initiation?
* Has he received an investigational drug during the 30 day period preceding study initiation? A yes answer to any of the above questions indicates that the individual is ineligible for enrollment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-07; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R. Pizarro,, M.D., Principal Investigator — SFBC Ft. Myers, Inc
Locations (1):
- SFBC Ft. Myers, Inc., Fort Myers, Florida, United States